CLINICAL TRIAL: NCT00588874
Title: Pilot Study to Assess the Skeletal Effects of Age-related Changes in Calcium and Vitamin D Metabolism in Men
Brief Title: Age Related Changes in Calciotropic Hormones and Their Impact on Male Osteoporosis
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Barbara I. Gulanski, MD, MPH, Yale University School of Medicine
Other Study IDs: 11946; Pepper Center Pilot Award
Record Dates: First submitted 2007-12-27; First posted 2008-01-09 (Estimated); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Low Bone Density
Keywords: male osteoporosis; male osteopenia; calciotropic hormones
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: men 50 yrs of age or older

SUMMARY:
The purpose of this pilot study is to generate preliminary data regarding the skeletal effects of age-related changes in calcium and vitamin D metabolism in older men.

ELIGIBILITY:
Inclusion Criteria:

* healthy men age 50 yrs and older

Exclusion Criteria:

* smokers
* known history of metabolic bone disease, known history of hypogonadism or renal insufficiency.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy men 50 yrs of age and older, without a known history of metabolic bone disease or renal insufficiency
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2000-10-01 (Actual); Primary Completion 2002-07-01 (Actual); Study Completion 2008-12-01 (Actual)

PRIMARY OUTCOMES:
Bone density of hip and spine | measured after screening evaluation

SECONDARY OUTCOMES:
calciotropic hormones, including calcium, PTH and vitamin D metabolites | measured after screening evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Barbara I Gulanski, MD, MPH, Principal Investigator — Yale University
Locations (1):
- Yale Center for Clinical Investigation, New Haven, Connecticut, United States